CLINICAL TRIAL: NCT02239081
Title: A Randomized, Double-blind, Single Ascending Dose, Safety, Tolerability, Pharmacokinetics Study of CTP-730 in Healthy Volunteers
Brief Title: A Safety and Tolerability Study of CTP-730 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Concert Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CP730.1001
Record Dates: First submitted 2014-09-09; First posted 2014-09-12 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Healthy
Keywords: Pharmacokinetics; Safety

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- CTP-730, 5 mg (Experimental): oral suspension, once daily.
  Interventions: Drug: CTP-730; Drug: Placebo for CTP-730
- CTP-730, 10 mg (Experimental): Oral Suspension, once daily.
  Interventions: Drug: CTP-730; Drug: Placebo for CTP-730
- CTP-730, 20 mg (Experimental): Oral Suspension, once daily.
  Interventions: Drug: CTP-730; Drug: Placebo for CTP-730
- CTP-730, 30 mg (Experimental): Oral Suspension, once daily.
  Interventions: Drug: CTP-730; Drug: Placebo for CTP-730
- CTP-730, 40 mg (Experimental): Oral Suspension, once daily.
  Interventions: Drug: CTP-730; Drug: Placebo for CTP-730
- CTP-730, 50 mg (Experimental): Oral Suspension, once daily.
  Interventions: Drug: CTP-730; Drug: Placebo for CTP-730
- CTP-730, 60 mg (Experimental): Oral Suspension, once daily.
  Interventions: Drug: CTP-730; Drug: Placebo for CTP-730

INTERVENTIONS:
Drug: CTP-730
Drug: Placebo for CTP-730

SUMMARY:
This is a Phase 1, single center, single-ascending dose, randomized study

DETAILED DESCRIPTION:
Following a Screening period of up to 21 days, eight (8) subjects in each cohort, 6 subjects randomized to CTP-730 and 2 subjects randomized to placebo, will be admitted to the clinical research unit (CRU) on the evening before dosing and remain sequestered at the study site until after the last inpatient blood sample is collected at 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteer subjects, 18 to 50 years of age, inclusive.

Exclusion Criteria:

* Current significant medical condition, laboratory abnormality, or psychiatric illness
* History of clinically significant central nervous system (eg, seizures), cardiac, pulmonary, metabolic, renal, hepatic, or gastrointestinal (GI) conditions
* PR interval ≥ 220 msec or QRS duration ≥ 120 msec or QTcB / QTcF interval > 450 msec
* Elevated liver function tests greater than twice the upper limit of normal
* Positive blood screen for human immunodeficiency virus (HIV antibody), hepatitis B virus surface antigen, or hepatitis C virus antibody
* Urinalysis positive for protein or glucose
* A positive screen for alcohol, drugs of abuse, or tobacco use.
* Inability to comply with food and beverage restrictions during study participation
* Donation or blood collection or acute loss of blood prior to screening

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2014-09; Primary Completion 2015-01 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Number and severity of adverse events | 3 days
Pharmacokinetics parameters | 96 hours
  Peak plasma concentration - Cmax by dose Area under the plasma concentration by time - AUC by dose

CONTACTS AND LOCATIONS:
Overall Officials: Ginny Braman, Study Director — Concert Pharmaceuticals, Inc.
Locations (1):
- CMAX, Adelaide, South Australia, Australia